CLINICAL TRIAL: NCT03356379
Title: Application de l'oxymétrie Dynamique Pour le Diagnostic Des pièges artériels poplités
Brief Title: Popliteal Artery Entrapment Syndrome & TRanscutaneoUS Oxymetry
Acronym: PETRUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2017-AO1887-46
Record Dates: First submitted 2017-11-22; First posted 2017-11-29 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Popliteal Entrapment Syndrome
Keywords: Diagnosis; Peripheral artery disease; sports
MeSH Terms: conditions — Popliteal Artery Entrapment Syndrome; Disease; Peripheral Arterial Disease | interventions — Blood Gas Monitoring, Transcutaneous

STUDY DESIGN:
Intervention Model Description: transcutaneous oximetry
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients (Experimental): Patients suspected of PES will have a transcutaneous oximetry test during tiptoeing
  Interventions: Diagnostic Test: Transcutaneous oximetry
- Controls (Sham Comparator): Healthy asymptomatic athletes will have a transcutaneous oximetry test during tiptoeing
  Interventions: Diagnostic Test: Transcutaneous oximetry

INTERVENTIONS:
Diagnostic Test: Transcutaneous oximetry — Measurement of TcpO2 on calves and chests. Calculation of the DROP index (decrease from rest of oxygen pressure)on both calves

SUMMARY:
Aim of the study is to test the feasibility of transcutaneous oxygen pressure (TcPO2) recording in the diagnosis of popliteal entrapment syndrome (PES) in 30 patients with suspected PES and 30 asymptomatic control heathy subjects

DETAILED DESCRIPTION:
Patients suspected of PES and healthy cpontrols after detailled explanation of the protocol will have a recording of tcpO2 on both calves and will perform a series of elevation on foot in the standing position.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Insurance company alffiliation Symptoms consistent with PES (patients) or absence of symptoms (controls)

Exclusion Criteria:

* Refuse to participate Exclusion period from another protocole

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-11-22 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Presence of a significant DROP decrease | 1 hour
  Comparison of DROP value between PES patients and controls

CONTACTS AND LOCATIONS:
Overall Officials: Pierre ABRAHAM, MD; PhD, Principal Investigator — University Hospital in Angers
Locations (1):
- CHU Angers, Angers, France

IPD SHARING:
Plan to Share IPD: Undecided